CLINICAL TRIAL: NCT02710682
Title: Ultrasound-guided Tendon Fenestration Versus Open Surgery for the Treatment of Chronic Lateral Epicondylosis of the Elbow: a Prospective, Randomized, Single Blind, Pilot Study.
Brief Title: Tendon Fenestration Versus Surgery for the Treatment of Chronic Lateral Epicondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE 15.327
Record Dates: First submitted 2016-03-08; First posted 2016-03-17 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2022-06

CONDITIONS: Epicondylitis of the Elbow; Tennis Elbow
Keywords: Lateral Epicondylitis of the elbow; Tendon Fenestration; Minimally invasive Surgery; Ultrasound-guided procedure; Ultrasonography; Elastography
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mini-open surgery (Active Comparator): Surgery
  Interventions: Procedure: Mini-open surgery
- Ultrasound-guided Tendon fenestration (Experimental): Tendon fenestration
  Interventions: Device: Ultrasound-guided Tendon fenestration

INTERVENTIONS:
Procedure: Mini-open surgery — This treatment will be administered by an orthopedic surgeon specialized in upper limb surgery.
  1. Skin disinfection; Local anesthesia (lidocaine 1%).
  2. Skin incision, slightly anterior to lateral epicondyle.
  3. Exposure of the plane between the tendon and fascia.
  4. Extensor Carpi Radialis Longus (ECRL) tendon is lifted to expose the Extensor Carpi Radialis Brevis (ECRB) tendon.
  5. Excision of diseased tissue of the ECRB tendon.
  6. ECRL tendon is sutured back to the fascia. The skin is closed.
  7. Patient is monitored for 30 minutes after procedure.
  Arms: Mini-open surgery
Device: Ultrasound-guided Tendon fenestration — This treatment will be administered by a fellowship-trained MSK radiologist.
  1. Patient's elbow at 70 degrees of flexion with the forearm pronated resting on an examination table.
  2. Skin disinfection. Local anesthesia, skin, superficial fascia and tendon, with lidocaine 1%.
  3. Using a 22 G needle under continuous ultrasound guidance, several passes (about 20-30) within the abnormal area of the tendon, contacting the bone, until the area softens.
  4. Patient monitored for 30 minutes, before being discharged.
  Arms: Ultrasound-guided Tendon fenestration

SUMMARY:
Lateral epicondylosis, also called tennis elbow or lateral epicondylitis, is a prevalent, painful syndrome of the elbow. It is refractory to conservative treatment measures, including rest, excentric and concentric exercises in approximately 20% of patients after 6 months. Corticosteroid injections can provide relief in the short term. Mini-open surgery may be proposed when the conservative treatment fails and studies have shown an efficacy of 70%. Ultrasound-guided tendon fenestration is a minimally-invasive technique which stimulates the physiological healing mechanisms of the tendon and appears promising for the treatment of chronic tendinopathies. To our knowledge, no studies have compared the US-guided fenestration technique to mini-open surgery for the treatment of chronic lateral epicondylosis.

The primary objective of this pilot study is to compare the efficacy of US-guided fenestration to mini-open surgery to reduce pain and improve functional status in workers suffering from chronic lateral epicondylosis refractory to 6-month conservative treatment.

This is a prospective single-blind randomized pilot study. Sixty-four subjects will be randomized into two intervention groups for treatment either by US-guided fenestration or mini-open surgery. The primary outcome of the study will be the Patient Rated Tennis Elbow Evaluation (PRTEE) score at 6 month post-procedure.

DETAILED DESCRIPTION:
STUDY DESIGN:

Phase II, prospective, two-arm, single-blind randomized controlled study.

SETTING:

Up to 64 patients (56 + 15% loss to follow-up) suffering from chronic lateral epicondylosis will be recruited by one of two orthopedists working in a specialized outpatient clinic, at the Centre Hospitalier de l'Université de Montréal (CHUM), a tertiary care academic center. Ultrasound examination of the elbow will be performed before the interventions.

RANDOMIZATION:

Using a computerized randomization list, the subjects will be randomized into the 2 treatment arms to be treated either by an US-guided tendon fenestration technique or by mini-open surgery. Randomization will be stratified by block sizes of 8.

FOLLOW UP Subjects' follow-up will extend over a period of 12 months - i.e., at 6 weeks and 3, 6 and 12 months post-intervention. The primary outcome will be the PRTEE score. Secondary outcomes will evaluate the impact of each procedure on: Pain-free grip (dynamometer), Medication Quantitative Scale, working activity (QuickDASH general and work modules; RA-WIS), Patient Global Impression of Change and Patient Satisfaction. The ultrasound examination will be repeated at 6 and 12 months. The predictive value of various B-mode parameters, color Doppler and elastography will be explored.

ANALYSIS:

The primary endpoint will be the proportion of subjects in each intervention arm presenting a reduction of at least 11/100 of the PRTEE score at 6 months post-intervention. The Fisher's exact test will be used to compare the proportion of subjects in each treatment group. The primary analysis will follow the intention-to-treat principle. Regarding the secondary endpoints, an ANOVA for repeated measures with two factors (time and group), a Fisher's exact test or a recursive partitioning analysis will be performed as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Workers
* Ability to read, understand and answer questionnaires in French or English
* Diagnosis of unilateral, lateral epicondylosis established by an orthopaedist, determined by clinical presentation and pain, ≥ 4/10 on a pain numerical rating scale, on palpation of the region slightly anterior and distal to the lateral epicondyle, exacerbated by the extension of the wrist or the middle finger when the elbow is in extension.
* Chronic epicondylosis, refractory to medical treatment conducted for at least six months, which includes rest and implementation of ergonomics to avoid soliciting the extensor tendons, and at least one of: physical therapy, a rehabilitation program with stretching and / or strengthening exercises, injection treatments (corticosteroids, autologous PRP) or extracorporeal shock waves.

Exclusion Criteria:

* Suspected tumor or infectious etiology
* Injection of corticosteroids during the last 3 months
* Hemorrhagic diathesis; anticoagulation (platelets <50,000, International Normalized Ratio (INR) > 2)
* Local infection
* History of elbow surgery or fracture
* History of inflammatory arthropathy
* Neck pain and radiculopathy
* Inability to provide informed consent because of a language problem, dementia or a major psychiatric disorder.

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Patient Rated Tennis Elbow Evaluation | Baseline and 6 months post-intervention
  Proportion of patients with a change of at least 11/100 points in the score of the Patient Rated Tennis Elbow Evaluation - 6 months

SECONDARY OUTCOMES:
Patient Rated Tennis Elbow Evaluation | Baseline and 6 weeks, 3 months, 12 months post-intervention
  Proportion of patients with a change of at least 11/100 points in the score over the time.
  Mean change in the score over the time.
QuickDASH main module | Baseline and 6 weeks, 3 months, 6 months and 12 months post-intervention
  Proportion of patients with a change of at least 8/100 points in the score over the time.
  Mean change in the score over the time.
QuickDASH Work module | Baseline and 6 weeks, 3 months, 6 months and 12 months post-intervention
  Proportion of patients with a change of at least 8/100 points in the score over the time.
  Mean change in the score over the time.
RA-WIS questionnaire | Baseline and 6 weeks, 3 months, 6 months and 12 months post-intervention
  Proportion of patients with score of at least 17 points over the time. Mean change in the score over the time.
Grip strength without pain | Baseline and 6 weeks, 3 months, 6 months and 12 months post-intervention
  Mean change over the time
Medication Quantitative Scale | 6 weeks, 3 months, 6 months and 12 months post-intervention
  Mean change over the time
Global Perception of Change | 6 weeks, 3 months, 6 months and 12 months post-intervention
  Proportion of patients reporting that their condition has significantly or moderately improved over the time
Level of satisfaction | 6 weeks, 3 months, 6 months and 12 months post-intervention
  Proportion of patients reporting that their condition has significantly or moderately satisfied over the time
Common Extensor Tendon Morphometric parameters measured at B-mode ultrasound | Baseline, 6 and 12 months post-intervention
  Recursive partitioning analysis
Common Extensor Tendon Elasticity measured at ultrasound elastography | Baseline, 6 and 12 months post-intervention
  Recursive partitioning analysis

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Bureau, MD, MSc, Principal Investigator — CRCHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lungu E, Grondin P, Tetreault P, Desmeules F, Cloutier G, Choiniere M, Bureau NJ. Ultrasound-guided tendon fenestration versus open-release surgery for the treatment of chronic lateral epicondylosis of the elbow: protocol for a prospective, randomised, single blinded study. BMJ Open. 2018 Jun 9;8(6):e021373. doi: 10.1136/bmjopen-2017-021373. PMID 29886446
- [Result] Bureau NJ, Tetreault P, Grondin P, Freire V, Desmeules F, Cloutier G, Julien AS, Choiniere M. Treatment of chronic lateral epicondylosis: a randomized trial comparing the efficacy of ultrasound-guided tendon dry needling and open-release surgery. Eur Radiol. 2022 Nov;32(11):7612-7622. doi: 10.1007/s00330-022-08794-4. Epub 2022 Apr 28. PMID 35482125
- [Result] Tobaly D, Tetreault P, Cloutier G, Choiniere M, Grondin P, Freire V, Julien AS, Bureau NJ. Assessing the treatment response of lateral elbow tendinopathy using time-dependent ultrasonography, Doppler imaging, and elastography. Insights Imaging. 2024 May 11;15(1):113. doi: 10.1186/s13244-024-01695-8. PMID 38734857